CLINICAL TRIAL: NCT00642694
Title: Time to Remission of Depressive Symptoms With Combined SSRI and Ramelteon
Acronym: TAKEDA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment discontinued based on mutually agreed upon decision by PI and funding sponsor
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Prabha Sunderajan, Clinical Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-031R; 112006-017
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Major Depressive Disorder; Insomnia
Keywords: MDD; Major Depressive Disorder; Depression; Initial Insomnia; sleep; difficulty sleeping; down; sad; Major Depressive Disorder(MDD) and initial insomnia
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders; Depression; Parasomnias | interventions — Escitalopram; ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Escitalopram tablets (starting dose of 10 mg with a maximum dose of 20 mg daily) + Ramelteon (One 8 mg capsule at night)
  Interventions: Drug: Escitalopram; Drug: Ramelteon
- 2 (Placebo Comparator): Escitalopram tablets (starting dose of 10 mg with a maximum dose of 20 mg daily) + Matching Placebo (One capsule at night)
  Interventions: Drug: Escitalopram; Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10 or 20mg qd based on symptoms at patient visit
  Other Names: Lexapro (escitalopram)
Drug: Ramelteon — Ramelteon 8 mg qd
  Other Names: Rozerem (Ramelteon)
  Arms: 1
Other: Placebo — Matching placebo qd
  Arms: 2

SUMMARY:
Hypothesis I: Patients in the SSRI + ramelteon treatment group will achieve remission (defined as an IDS-C30 score of 11 or less) more quickly than those in the SSRI + placebo group.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the time to remission in depression with initial insomnia using the SSRI antidepressant escitalopram combined with ramelteon or placebo. Patients will be assessed at each visit for depressive symptoms and insomnia, using the 30-item Inventory of Depressive Symptoms, Clinician-Rated version (IDS-C30; Rush et al 1986; Rush et al., 1996) as the primary outcome measure. The IDS self-report version will be used to assess self-reported changes in symptom severity. The 17 item Hamilton Rating Scale for Depression, (HRSD17; Hamilton, 1960) will also be administered, as it is the most commonly utilized depression symptom severity measure at this time.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent.
* Primary diagnosis of MDD with initial insomnia.
* Age 18-70.
* Screening HRSD17 score greater than or equal to 16 or CGI-S score of at least 4.
* Subjective report of difficulties with initial insomnia with a score of 2 or greater on the IDS-C30 item addressing this symptom (#1). Middle and late insomnia may also be present so long as initial insomnia is present.

Exclusion Criteria:

* Presence of significant comorbid medical condition based on laboratory test, physician information, or evidence at examination; this includes severe sleep apnea, seizure disorder, or chronic obstructive pulmonary disease (COPD).
* Patient report or evidence (based on physical examination or laboratory tests) of significant medical abnormalities; this includes severe sleep apnea, seizure disorder, or COPD.
* Presence of other psychological disorders, including depression due to other comorbid conditions, currently suicidal or high suicide risk, current or past psychotic disorders of any type, bipolar disorder (I, II, or NOS), schizophrenia, or schizoaffective disorder, anorexia, bulimia, obsessive compulsive disorder, alcohol or substance abuse within the last 6 months, or patients with comorbid psychiatric conditions that are relative or absolute contraindications to the use of escitalopram or ramelteon.
* Concomitant (i.e. within 2 weeks; 4 weeks for fluoxetine or MAOIs) pharmacological or psychotherapeutic treatment including but not limited to anxiolytics, neuroleptics, mood stabilizers, sleep aids including over the counter melatonin, and/or other agents without proven antidepressant efficacy, cognitive behavioral therapy; current use of other medications that would be contraindicated with ramelteon or escitalopram,, as determined by the study doctor.
* Failure to respond to 2 adequate courses of SSRI class antidepressant in the current episode (as measured by the Antidepressant Treatment History Form).
* Hospitalization for mental illness within the past year.
* For women, currently pregnant, planning to become pregnant in the next year, or breastfeeding.
* Patient does not speak English. (Patient needs to be fluent in written and oral English because not all assessments are available and/or validated in languages other than English).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- See also: Mood Disorders Research Program and Clinic — http://www.utsouthwestern.edu/utsw/home/.research/depression

RESULTS

PARTICIPANT FLOW:
Groups:
- Escitalopram + Ramelteon: active augmentation
- Escitalopram + Placebo: Placebo augmentation
Period: Overall Study
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Started | 14 | 15
Completed | 8 | 11
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (12.4) | 42.0 (11.4) | 42.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Remitters on IDS-C30 at Week 12
Description: Remission as defined by a score of <12 on the Inventory of Depressive Symptomatology, Clinician-Rated version (IDS-C30) at Week 12; minimum possible score = 0, maximum possible score = 84; higher scores indicate worse symptom severity
Time Frame: 12 Weeks
Population: Participants who were randomized to treatment and completed Week 12 were included in analyses
Measure: Number; unit: percentage of participants
Groups:
- Escitalopram + Placebo: control group
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 10 | 11
percentage of participants | 20 | 36
Statistical Analysis 1: Comparison: Escitalopram + Ramelteon vs Escitalopram + Placebo; Test type: Superiority; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Sleep Latency
Description: Number of minutes until fell asleep
Time Frame: 12 weeks
Population: Number of Participants with analyzable data for this outcome measure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 13 | 15
minutes | 30.4 (29.1) | 15.8 (16.2)

3. Secondary Outcome: Short-Form Health Survey - Version 2 (SF-36)
Description: The Short-Form Health Survey - version 2 (SF-36) is a self-report inventory measuring different domains of health-related quality of life: Physical Functioning, Physical Role Functioning, Bodily Pain, General Health, Vitality, Social Functioning, Emotional Role Functioning, and Mental Health. Scores range from 0 to 100, with higher scores indicating better perceived health and functioning.
Time Frame: 12 Weeks
Population: Please note that the study was terminated early and may be underpowered to perform these analyses; results should be interpreted with caution.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 14 | 15
score on a scale
  Physical Functioning | 80.50 (28.43) | 88.33 (16.42)
  Social Functioning | 69.44 (37.56) | 68.75 (27.95)
  Physical Role Functioning | 75.00 (28.93) | 86.11 (17.89)
  Emotional Role Functioning | 67.59 (24.45) | 75.00 (20.10)
  Mental Health | 68.00 (25.30) | 70.42 (21.16)
  Vitality | 49.38 (27.55) | 54.69 (20.49)
  Bodily Pain | 75.31 (25.93) | 87.96 (19.22)
  General Health | 74.90 (21.12) | 79.25 (20.23)

4. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) measures satisfaction and enjoyment in various domains of functioning: physical health, feelings, work, household duties, school/course work, leisure time activities, social relations, and general activities. The raw score is converted into a percent of the maximum possible score and ranges from 0 to 100. Higher scores indicate greater enjoyment and satisfaction.
Time Frame: 12 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 14 | 15
score on a scale | 69.84 (14.44) | 70.24 (12.27)

5. Secondary Outcome: Social Adjustment Scale - Self-Report (SAS-SR)
Description: The Social Adjustment Scale - Self-Report (SAS-SR) is a 54-item self-report measure of instrumental and expressive role performance. Each item is rated on a 5-point scale, and a mean item score (ranging from 1-5) is obtained, with higher scores indicating greater impairment.
Time Frame: 12 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mean score on a scale
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 14 | 15
mean score on a scale | 2.09 (0.39) | 2.03 (0.46)

6. Secondary Outcome: Work and Social Adjustment Scale (WSAS)
Description: The Work and Social Adjustment Scale (WSAS) is 5-item self-report measure designed to identify functional impairment that is attributed to an identified problem or condition. and has been used in studies of depression and anxiety. Scores range between 0-40, with higher scores indicating worse functioning.
Time Frame: 12 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 14 | 15
score on a scale | 15.56 (11.42) | 13.91 (12.89)

7. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire (WPAI)
Description: The Work Productivity and Activity Impairment Questionnaire (WPAI) was used to report impairment while working or performing usual daily activities as a result of health problems. The activity impairment item (#6 of WPAI) is rated on a scale of 0-10, with higher scores indicating greater impairment. Scores are multiplied by 10 to obtain percent impairment.
Time Frame: 12 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of time activity was impaired
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 14 | 15
percentage of time activity was impaired | 40.00 (35.36) | 32.50 (27.34)

8. Secondary Outcome: Patient Perception of Benefits of Care (PPBC)
Description: The Patient Perception of Benefits of Care (PPBC) assesses how much patients believe their quality of life will improve in response to medical care or treatment. Scores range between 10-50, with lower scores indicating greater belief that treatment will improve quality of life.
Time Frame: 12 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 14 | 15
score on a scale | 20.33 (8.38) | 20.08 (12.50)

9. Secondary Outcome: Hamilton Rating Scale for Depression 17-item
Description: The Hamilton Rating Scale for Depression is a clinician-administered rating scale that assesses severity of depressive symptoms and is one of the most widely used and validated symptom severity measures for depression. Each of the 17 items is rated by the clinician on either a 3- or a 5 point scale. Total scores range from 0-52, with higher scores indicating greater depressive symptoms.
Time Frame: 12 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Number analyzed (Participants) | 14 | 15
score on a scale | 8.33 (6.26) | 10.08 (6.36)

ADVERSE EVENTS:
Time Frame: During 12 weeks of active treatment, plus time between consent and treatment and 2-weeks post-treatment
Arm/Group | Escitalopram + Ramelteon | Escitalopram + Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 13/14 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram + Ramelteon (N=14) | Escitalopram + Placebo (N=15)
constipation (Gastrointestinal disorders) | 3 (5) | 2 (2)
vivid dreams (Nervous system disorders) | 0 (0) | 1 (1)
pain and discomfort in genital area (Reproductive system and breast disorders) | 0 (0) | 1 (1)
sinus headache (Nervous system disorders) | 1 (1) | 1 (1)
palpitations (Cardiac disorders) | 1 (1) | 2 (3)
tiredness (General disorders) | 4 (12) | 1 (1)
insomnia (Nervous system disorders) | 1 (1) | 0 (0)
heartburn/indigestion/dyspepsia (Gastrointestinal disorders) | 1 (2) | 3 (3)
headache (Nervous system disorders) | 7 (13) | 5 (15)
dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (10)
stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
muscle and joint aches and pains (Musculoskeletal and connective tissue disorders) | 5 (15) | 2 (2)
increased appetite (Gastrointestinal disorders) | 1 (1) | 1 (1)
weight gain (Gastrointestinal disorders) | 1 (1) | 0 (0)
metallic taste (Nervous system disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (7) | 5 (5)
altered taste (Nervous system disorders) | 1 (3) | 0 (0)
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (3)
toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
tingling (Nervous system disorders) | 0 (0) | 1 (1)
head fullness (Nervous system disorders) | 0 (0) | 1 (2)
fidgetiness/restlesness (Nervous system disorders) | 1 (1) | 3 (12)
increased urination (Renal and urinary disorders) | 1 (2) | 0 (0)
stomach cramps (Gastrointestinal disorders) | 1 (4) | 0 (0)
swollen lymph node (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
increased yawning (General disorders) | 0 (0) | 2 (5)
erectile dysfunction (Reproductive system and breast disorders) | 2 (6) | 0 (0)
sinus infection/allergy (General disorders) | 2 (3) | 0 (0)
increased perspiration (General disorders) | 1 (1) | 0 (0)
dizziness (General disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
decreased libido (Reproductive system and breast disorders) | 0 (0) | 2 (6)
pulled back muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hot flashes (Reproductive system and breast disorders) | 0 (0) | 1 (3)
blurred vision (Eye disorders) | 0 (0) | 1 (1)
heart pounding (Cardiac disorders) | 0 (0) | 1 (1)
increased anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chills (General disorders) | 1 (1) | 0 (0)
fever (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No